CLINICAL TRIAL: NCT07024940
Title: Acute Effects of Coffee, Anthocyanin-Caffeine Supplement and Placebo on Exercise Performance Markers
Brief Title: Short-term Effects of Caffeine and a Multi-ingredient Pre-workout on Exercise Performance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Hossein Rafiei, Assistant Professor, Nutrition and Dietetics, St. Louis University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 34611
Record Dates: First submitted 2025-06-02; First posted 2025-06-17 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-06

CONDITIONS: Coffee; Anthocyanins; Exercise Performance
Keywords: Coffee; Caffeine; Wingate; Anthocyanin-Caffeine; 1-mile; VO2 max; pre-workout; supplement
MeSH Terms: interventions — Dietary Supplements; Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ethiopian Coffee (Experimental): A light roast Ethiopian Coffee is used based on previous research using the same technique for brewing. The coffee is brewed using the Aeropress coffee maker and the Timemore C3Pro hand grinder to grind the coffee. The recipe uses 15 grams of ground coffee set at the same grind setting (16 clicks) and 200 grams of water to have a target cup size of 175 mL plus 50 grams of ice to rapidly cool down the drink for consumption.
  Interventions: Other: Ethiopian Coffee
- Anthocyanin-Caffeine (Experimental): An anthocyanin-caffeine pre-workout supplement containing 120 mg of anthocyanins from New Zealand Blackcurrant berries, along with 120 mg of caffeine. This single-serve packet is stirred into 8 ounces of water and served.
  Interventions: Dietary Supplement: Supplement
- Water (Placebo Comparator): Water used as a constant water intake across all three arms
  Interventions: Other: Water (Placebo)

INTERVENTIONS:
Other: Ethiopian Coffee — Ethiopian Coffee is used as a real-world example of one of the most common drinks in the world.
  Arms: Ethiopian Coffee
Dietary Supplement: Supplement — A pre-workout supplement that contains anthocyanins and caffeine as ergogenic aids
  Arms: Anthocyanin-Caffeine
Other: Water (Placebo) — Bottled water acting as the placebo
  Arms: Water

SUMMARY:
The investigators are conducting a study to see how a commercial pre-workout supplement, coffee, and water affect how well people perform. The study is conducted across four visits. The first visit is to assess the participants, and the next three visits are for testing. Each participant will drink a randomly assigned beverage 45 minutes before testing. Throughout the study, the participants will complete three testing days-each at least three days apart-so they can try all three drinks. The first test is the Wingate test, where the participants pedal as fast as they can for 30 seconds against a set resistance. The second test is a 1-mile treadmill run/walk on an incline, where the participant tries to complete the distance as fast as possible. The third test measures reaction time using light-up buttons to see how quickly a participant responds by touching them. These tests will help determine if any of the drinks improve performance. The results can help people choose the best drink for their workouts or races.

DETAILED DESCRIPTION:
This study is being conducted to evaluate how a commercial pre-workout supplement with multiple ingredients and coffee affects how people perform during exercise testing. The study takes place over 4 separate lab visits. The first lab visit is an assessment for each participant to help define the population to be tested. Then, three testing visits will be identical in design but will differ in the intervention given to the participant. Each participant will consume the pre-workout, coffee, and a placebo in a randomized order. At the beginning of each visit, the participant will consume their assigned beverage. The participants will then start a warm-up after 30 minutes of consuming the assigned beverage. After the 10-minute warm-up, the participant will rest for five minutes before conducting the testing. In the testing visits, participants will conduct a 1-mile treadmill run, in which the participant will determine their speed using a 1% incline. This allows the participant to control the speed, allowing them to try as hard as they can. The next test will be a Wingate cycle ergometer test. The test contains a 20-second warm-up followed by a three-second period where the participant will pedal as fast as they can until the test begins, then they will do an all-out effort for 30 seconds. The participant will then conduct an agility reaction time test to measure any benefits the interventions may have on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy male or female adult aged 18-35 years old
* Regularly engaged in resistance training or aerobic exercise at least 3 times per week, at least 30 minutes a week for the past 6 months
* Able to provide written informed consent

Exclusion Criteria:

* Have a history of or currently have a cardiovascular or metabolic disease (e.g., diabetes, prediabetes, hypertension, arrhythmia, heart attack, stroke, non-alcoholic fatty liver disease, chronic kidney disease)
* History of seizure disorder
* Currently taking prescription medications (e.g., beta-blockers, antidepressants, anti-anxiety, pain killers)
* Currently pregnant, breastfeeding, pregnant within the past year, or a chance of being pregnant
* Recent participation in another clinical trial
* Any sensitivities to caffeine, coffee, berries, maltodextrin, monk fruit extract, or any known food allergies
* Currently undertaking serious exercise training (6 or more days of the week)
* Recently started taking creatine or beta-alanine daily within the past 3 months. (If greater than 3 months taken consistently is okay)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-25 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in anaerobic power measured by a 30-second all-out effort on a cycle ergometer | At 45 minutes post-dose for each intervention condition
  The primary outcome measured is the change in anaerobic power measured by a 30-second all-out effort on a cycle ergometer using the Wingate testing. This test will determine whether the interventions confer any performance benefit compared to the placebo.

SECONDARY OUTCOMES:
1-mile Treadmill time trial | At 45 minutes post-dose for each intervention condition
  The 1-mile treadmill time trial will help determine if either of the interventions allows for a faster time, translating to an increase in physical performance.
Agility Reaction Time | At 45 minutes post-dose for each intervention condition
  Agility reaction time will be measured with light-up buttons, where participants will need to touch the light to measure time. This test will identify if either intervention can reduce reaction time, which may reflect improvements in neuromotor performance.

CONTACTS AND LOCATIONS:
Overall Officials: Hossein Rafiei, PhD, Principal Investigator — St. Louis University
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castañeda-Babarro A. The Wingate Anaerobic Test, a Narrative Review of the Protocol Variables That Affect the Results Obtained. Applied Sciences. 2021; 11(16):7417. https://doi.org/10.3390/app11167417
- [Background] Lindsey ZR, Williams JR, Burgess JS, Moore NT, Splichal PM. Caffeine content in filter coffee brews as a function of degree of roast and extraction yield. Sci Rep. 2024 Nov 25;14(1):29126. doi: 10.1038/s41598-024-80385-3. PMID 39582028
- [Background] Jardine WT, Aisbett B, Kelly MK, Burke LM, Ross ML, Condo D, Periard JD, Carr AJ. The Effect of Pre-Exercise Hyperhydration on Exercise Performance, Physiological Outcomes and Gastrointestinal Symptoms: A Systematic Review. Sports Med. 2023 Nov;53(11):2111-2134. doi: 10.1007/s40279-023-01885-2. Epub 2023 Jul 25. PMID 37490269
- [Background] Peacock OJ, Thompson D, Stokes KA. Voluntary drinking behaviour, fluid balance and psychological affect when ingesting water or a carbohydrate-electrolyte solution during exercise. Appetite. 2012 Feb;58(1):56-63. doi: 10.1016/j.appet.2011.08.023. Epub 2011 Sep 29. PMID 21986184
- [Background] Lee JD, Sterrett LE, Guth LM, Konopka AR, Mahon AD. The effect of pre-exercise carbohydrate supplementation on anaerobic exercise performance in adolescent males. Pediatr Exerc Sci. 2011 Aug;23(3):344-54. doi: 10.1123/pes.23.3.344. PMID 21881155
- [Background] Kaczka P, Batra A, Kubicka K, Maciejczyk M, Rzeszutko-Belzowska A, Pezdan-Sliz I, Michalowska-Sawczyn M, Przydzial M, Plonka A, Cieszczyk P, Huminska-Lisowska K, Zajac T. Effects of Pre-Workout Multi-Ingredient Supplement on Anaerobic Performance: Randomized Double-Blind Crossover Study. Int J Environ Res Public Health. 2020 Nov 9;17(21):8262. doi: 10.3390/ijerph17218262. PMID 33182295
- [Background] Krzysztof, Wioleta Dorobek, Katarzyna Stankiewicz, Janusz Świeczkowski-Feiz. The Role of Caffeine in Enhancing Physical Performance: From Metabolism to Muscle Function. Journal of Education, Health and Sport. 2024;59. doi:10.12775/JEHS.2024.59.010